

Sponsor Name: Sound Pharmaceuticals, Inc.

Statistical Analysis Plan Version No.: Final 1.0

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

| STATISTICAL ANALYSIS PLAN | |
|---|---|
| Study Title:s | A Phase 2b, randomized, double-blind, placebo-controlled study to |
| | evaluate the safety and efficacy of SPI-1005 in Meniere's disease |
| Sponsor Identification: | Sound Pharmaceuticals, Inc. |
| Phase: | Phase 2b |
| Sponsor Study Number: | SPI-1005-251 |
| EA Study Number: | SPI-1005-251 |
| Responsible Biostatistician: | Prabhu S |
| Responsible Biostatistician. | Lead Biostatistician |
| | Ecron Acunova Limited |
| | Mobius Towers,SJR i-Park |
| | EPIP, Whitefield, |
| | Bangalore – 560 066 |
| | E-mail: <u>Prabhu.Siva@navitaslifesciences.com</u> |
| Date of SAP: | 30MAY2019 |
| Version: | Final 1.0 |
| Scope: | Final |

**NCT Number:** 03325790

# **ECRON ACUNOVA**

Statistical Analysis Plan

Version No.: Final 1.0

Sponsor Study No: SPI-1005-251

Sponsor Name: Sound Pharmaceuticals, Inc.

NLS Study Code: SPI -1005 -251

Short Title of Study: SPI -1005 -251 (Sound Pharmaceuticals, Inc)

#### **SIGNATURES**

Prepared by:

Riya Goel

Associate Biostatistics

Biostatistics & Programming

Ecron Acunova Ltd.

Bangalore, India

Signature


30 MAY 2019 Date (DD/MMM/YYYY)

Reviewed by:

Prabhu S

Lead Biostatistician

Biostatistics & Programming

Ecron Acunova Ltd.

Bangalore, India

(3.9)

30 MAY 2019

Signature

Date (DD/MMM/YYYY)

#### Approved by:

Jonathan Kil, MD Chief Medical Officer Sound Pharmaceuticals, Inc. 4010 Stone Way North Suite 120

Seattle, WA 98103

Jonathan Kil, MD

nathan Kii, MD

Jordathan Kil (May 30, 2012)

Signature

30May2019

Date (DD/MMM/YYYY)

#### Confidentiality Statement

This document is confidential and proprietary to Sponsor and EA and for restricted circulation and access only. No part of it may be transmitted, reproduced, published or used by any person/s without prior written authorization.



Sponsor Study No: SPI-1005-251

 Sponsor Name: Sound Pharmaceuticals, Inc. Version No.: Final 1.0

NLS Study Code: SPI-1005-251

Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

# TABLE OF CONTENTS

| SIGN | NATURES | | 2 |
|------|----------------|-----------------------------------------------|----|
| TAB | LE OF CONT | TENTS | 3 |
| 1 | DOCUMEN | T HISTORY | 5 |
| 2 | ABBREVIA | TIONS | 6 |
| 3 | DOCUMEN | TS | 8 |
| 4 | INTRODUC | CTION | 8 |
| 5 | STUDY OB. | JECTIVES | 8 |
| - | 5.1Primary ( | Objectives | 8 |
| | 5.2Secondar | | 9 |
| 6 | STUDY DE | SIGN | 9 |
| | 6.10verview | <b>y</b> | 9 |
| | 6.2Paramete | | 11 |
| | 6.2.1 | Primary Parameter | |
| | 6.2.2 | Secondary Parameters | 12 |
| | 6.2.3 | Safety Parameters | |
| | 6.2.4 | Exploratory Parameters | 12 |
| 7 | GENERAL S | STATISTICAL CONSIDERATIONS | 12 |
| | 7.1Description | ve Statistics | 12 |
| | 7.2Randomiz | zation and Blinding Process | 13 |
| | 7.3 Analysis | | 14 |
| | 7.3.1 | Randomized Population | 14 |
| | 7.3.2 | Intent-to-Treat (ITT) Analysis Population | |
| | 7.3.3 | Safety Analysis Population | |
| | 7.3.4 | Per-Protocol Population | |
| | 7.3.5 | PK Analysis Population | |
| | 7.4Protocol | | 15 |
| | 7.5Data Han | dling | 15 |
| | 7.5.1 | Imputation of Missing data | 15 |
| | 7.6Sample S | Size Calculation | 15 |
| | 7.7Interim A | | 15 |
| | | ns and Derived Variables | 16 |
| | 7.9Statistical | 1 Software | 17 |
| 8 | STATISTIC | AL ANALYSES | 17 |
| | 8.1.1 | Subject Disposition | 17 |
| | 8.1.2 | Inclusion/Exclusion Criteria | 17 |
| | 8.1.3 | Demographic Data and Baseline Characteristics | 18 |
| | 8.1.4 | Medical History | |
| | 8.1.5 | Prior and Concomitant Medication | 18 |
| | 8.2Extent of | Exposure and Compliance | 19 |
| | 8.2.1 | Treatment Exposure | 19 |

# **Confidentiality Statement**

This document is confidential and proprietary to Sponsor and EA and for restricted circulation and access only. No part of it may be transmitted, reproduced, published or used by any person/s without prior written authorization. 5



Statistical Analysis Plan Version No.: Final 1.0


Sponsor Study No: SPI-1005-251

Sponsor Name: Sound Pharmaceuticals, Inc.

| NLS | NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceutical | | Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, In | ls, Inc) |
|---|---|---|---|---|
| | 8.2.2 | Treatment Compliance | | 19 |
| | 8.3Efficacy | Analysis | | 19 |
| | 8.3.1 | Analysis of Primary Endpo | oint | 19 |
| | 8.4Safety Aı | | | 23 |
| | | | ations | |
| | 8.4.3 | | | |
| | 8.4.4 | • | | |
| | | okinetic Analysis | | 25 |
| | 8.6Multicen | | | 26 |
| | 8.7Subgroup | Analyses | | 26 |
| 9 | <b>DEVIATIO</b> | N FROM THE STUDY PRO | OTOCOL | 27 |
| | 9.1.1 | Exploratory Analysis | | 28 |
| 10 | SOPS FOR | ANALYSIS AND REPORT | ING | 29 |
| 11 | DATABASI | E LOCK AND UNBLINDIN | IG | 29 |
| 12 | REFERENC | CES | | 30 |
| 13 | LIST OF RE | EPORTED TABLES | | 31 |
| 14 | LIST OF RE | EPORTED FIGURES | | 36 |
| 15 | LIST OF RE | EPORTED SUBJECT DATA | LISTINGS | 38 |



Version No.: Final 1.0  Sponsor Name: Sound Pharmaceuticals, Inc.

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

# **1 DOCUMENT HISTORY**

| Version | Date | Change to previous version |
|-----------|-----------|----------------------------|
| Final 1.0 | 30MAY2019 | Nil |




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

# **2** ABBREVIATIONS

| ABBREVIATIONS | DEFINITION |
|---|---|
| AE | Adverse Event |
| AE(DAE) | Discontinuation of the study due to Adverse Events |
| ATC | Anatomical Therapeutic Chemical Classification |
| AUC <sub>0-t</sub> | Area under the curve time 0 to time t |
| Bid | Twice-daily dosing |
| BMI | Body Mass Index |
| CBC | Complete Blood Count |
| CFR | Code of Federal Regulations |
| C <sub>max</sub> | Maximum concentration |
| CRF | Case Report Form |
| CRO | Contract Research Organization |
| CV | Coefficient of Variation |
| dB | decibel, 1/10th of a Bel—measure of ratios on a logscale |
| dBHL | dB Hearing Level |
| EXP | Exponential |
| GCP | Good Clinical Practice |
| G.Mean | Geometric Mean |
| Hz | Hertz—unit of measure for frequency |
| IQR | Inter Quartile Range |
| ICH | International Conference on Harmonization |
| LCMS | Liquid Chromatography-Mass Spectrometry |
| mg | milligram |
| MD | Meniere's disease |
| MedDRA | Medical Dictionary for Regulatory Activities |
| Max | Maximum |
| Min | Minimum |
| NA | Not Applicable |
| PI | Principal Investigator |
| PK | Pharmacokinetics |



Statistical Analysis Plan

Sponsor Name: Sound Pharmaceuticals, Inc. Version No.: Final 1.0 

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

| Po | By mouth |
|------|-----------------------------|
| PTA | Pure-Tone Audiometry |
| Q1 | First Quartile |
| Q3 | Third Quartile |
| SAE | Serious Adverse Event |
| SAS | Statistical Analysis System |
| SD | Standard Deviation |
| SIC | Subject Identification Code |
| SNR | Signal-to-Noise Ratio |
| SPI | Sound Pharmaceuticals, Inc. |
| SQRT | Square Root |
| TFI | Tinnitus Functional Index |
| TL | Tinnitus Loudness |
| TTS | Temporary Threshold Shift |
| VSS | Vertigo Symptoms Scale |
| WINT | Words-in-Noise Test |




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### 3 DOCUMENTS

This statistical analysis plan is based on the study protocol SPI-1005-251, version 1.00 dated 21AUG2017.

### 4 INTRODUCTION

This Statistical Analysis Plan (SAP) is based on the relevant sections of study protocol and includes also the Tables, Listings and Figures (TLF) Specifications. The purpose of the SAP is to describe in more detail how the analyses are to be performed and presented. It quotes the relevant statements directly from the protocol, but it does not give a full description of study design etc.

The TLF Specifications specify the output to support the analysis. The TLF Specifications are considered as a guideline for producing the output.

The SAP will be finalized prior to database lock or any unblinding of study team members.

The objectives of this Phase 2b, randomized, double-blind, Placebo-controlled study are to demonstrate the safety and efficacy of SPI-1005 for the treatment of Meniere's disease.

### **5** STUDY OBJECTIVES

### 5.1 Primary Objectives

- > To determine the Safety of SPI-1005 treatment in adults with Meniere's disease.
- To determine the Efficacy of SPI-1005 with the following clinically validated methods and measures (responder analysis):
  - Primary pure-tone audiometry assessment (250, 500 or 1000 Hz): Improvements from baseline of ≥10 dB at 1 frequency
  - Secondary pure-tone audiometry assessments (250, 500 or 1000 Hz): Improvements from baseline of ≥10 dB at 2 adjacent frequencies or ≥20 dB at 1 frequency
  - Primary Words-in-Noise Test assessment (0-35): Improvements from baseline of ≥10%
  - Secondary Words-in-Noise Test assessments (0-35): Improvements from baseline of ≥20% or ≥4 words
  - Tinnitus Functional Index (TFI):  $(0-100) \ge 10$  pt. reduction from baseline
  - Tinnitus Loudness: Q#2 of TFI:  $(0-10) \ge 2$  pt. reduction from baseline
  - Vertigo Symptom Scale (0-60):  $\geq 6$  pt. reduction from baseline

The responder analysis from each method and measure will be compared between treatment groups for significance.

- The efficacy of SPI-1005 treatment in adults with Meniere's disease will be based on:
  - ➤ Improvement in sensorineural hearing loss using pure-tone audiometry at 250, 500, or 1000 Hz; or



Sponsor Name: Sound Pharmaceuticals, Inc.

Version No.: Final 1.0 

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

Word recognition score using WINT at 24, 20,16, 12, 8, 4 and 0 SNR; or

> Improvement in the Tinnitus Functional Index (TFI); or

> Improvement in Tinnitus Loudness (TL); or

➤ Improvement in the Vertigo Symptoms Scale (VSS)

#### 5.2 Secondary Objectives

Statistical Analysis Plan

To determine the pharmacokinetics at each dosing level of SPI-1005.

# **6** STUDY DESIGN

#### 6.1 Overview

This clinical trial is a phase 2b, randomized, double-blind, placebo-controlled study to evaluate the safety and efficacy of SPI-1005 in Meniere's disease. The study is planned to be conducted in adult volunteers with Meniere's Disease (probable or definitive diagnosis) with active symptoms in the months preceding study enrollment. Study participants will be randomized into three dosing arms: SPI-1005 200 mg/BID, SPI-1005 400 mg/BID, or placebo (1:1:1). This double-blind study will evaluate both safety and efficacy of the investigational treatment.

Participants aged 18-75 years, with probable or definitive Meniere's disease will undergo baseline testing to assess severity of sensorineural hearing loss, tinnitus and vertigo. This is a multicenter study that includes patients from approximately 12 US sites.

During the study, and 28 days after completion of treatment, participants will be evaluated for safety (adverse events, physical examinations, vital signs and clinical laboratory testing (CBC, serum chemistry). Trough plasma levels of ebselen and its major metabolite (2-glucuronyl selenobenzanilide) will be evaluated using liquid chromatography-mass spectrometry (LCMS) at specified visits. Additionally, plasma will be analyzed for selenium at the corresponding visits. Female participants will receive pregnancy testing at visit 1, and those found to be pregnant will be excluded from the study and monitored for adverse events.

The effect of SPI-1005 on hearing and balance will be evaluated. Hearing will be evaluated at baseline, at the end of 28 days of study treatment, and 28 days after completing study treatment.

Tinnitus and vertigo will be evaluated with the Tinnitus Functional Index (TFI) and the Vertigo Symptoms Scale (VSS), respectively. These tests will be administered at baseline, on days 14 and 28




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

of treatment, and 28 days after treatment. Hearing thresholds (HL) will be determined using pure-tone audiometric (air conduction) testing at 250, 500, 1000, 2000, 3000, 4000, 6000, and 8000 Hz, bilaterally. In addition, bone conduction testing with masking will be conducted if the air conduction threshold is >15 dBHL at 250, 500, 1000, 2000, or 4000 Hz. Bone conduction testing will only be performed at screening and in the affected ear (>15 dBHL). A word recognition test using the Wordsin-Noise Test (WINT) at 24, 20, 16, 12, 8, 4, and 0 Signal-to-Noise ratio (SNR) will be used to evaluate hearing.

Following completion of informed consent process and baseline assessments, the study participants will be evaluated by the investigator for enrollment eligibility. Participants that meet enrollment criteria will be randomized and assigned a Subject Identification Code from the list of Subject Identification Codes. The Subject Identification Code must be carefully matched to the study drug before the study drug is dispensed at Clinic Visits 1, and 2.

A general diagram of the study design is provided in Figure 1.



Statistical Analysis Plan


NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)



#### 6.2 Parameters

All parameters through which the study objectives will be carried out, should be listed. Exact computations will be declared in section 7.8 Definitions and Derived Variables.

# 6.2.1 Primary Parameter

- ➤ Efficacy of SPI-1005 will be determined by the following clinically significant methods and measures (responder analysis):
- ➤ Pure-tone audiometry assessment (250, 500 or 1000 Hz): Improvements from baseline of ≥10 dB at 1 frequency
- ▶ Words-in-Noise Test assessment (0-35): Improvements from baseline of  $\geq$ 10%
  - Tinnitus Functional Index (TFI)  $(0-100) \ge 10$  pt. reduction from baseline

# **Confidentiality Statement**

This document is confidential and proprietary to Sponsor and EA and for restricted circulation and access only. No part of it may be transmitted, reproduced, published or used by any person/s without prior written authorization.




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

■ Tinnitus Loudness: Q#2 of TFI  $(0-10) \ge 2$  pt. reduction from baseline

• Vertigo Symptom Scale  $(0-60) \ge 6$  pt. reduction from baseline

#### **6.2.2** Secondary Parameters

Pharmacokinetics parameters will be analyzed for the following parameters:

- 1.  $AUC_{0-t}$  (mg h/L)
- 2.  $C_{max}$  (mg/L)

#### **6.2.3** Safety Parameters

- > Safety of SPI-1005 treatment in adults with Meniere's disease will be analysed using:
  - Physical examinations
  - Vital signs
  - Adverse events
  - Hematology (CBC)
  - Serum chemistries.

### **6.2.4** Exploratory Parameters

- Secondary pure-tone audiometry assessments (250, 500 or 1000 Hz): Improvements from baseline of ≥10 dB at 2 adjacent frequencies or ≥20 dB at 1 frequency
- Secondary Words-in-Noise Test assessments (0-35): Improvements from baseline of ≥20% or ≥4 words

### 7 GENERAL STATISTICAL CONSIDERATIONS

#### 7.1 Descriptive Statistics

The following descriptive statistics will be calculated for continuously distributed data:

- r
- Mean
- Standard Deviation (also denoted as SD)
- Minimum (also denoted as Min)
- Median
- Maximum (also denoted as Max)
- Inter Quartile Range (IQR)




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

For categorical variables, counts and percentages will be calculated.

For continuous variables, the decimal places for n, minimum and maximum will be provided as per the reported value. Decimal places for mean, Q1, Q3 and median will be reported one decimal place more than the reported value. The decimal place for standard deviation will be reported two decimal places more than the reported value.

In all statistical tables, p-values will be reported as specified by the statistical program used, at least up to three decimal places. P-values less than 0.001 will be reported as provided by SAS®, Version 9.2 or higher (e.g. '<0.0001'). All tests will be two-sided at the  $\alpha$  = 0.05 level of significance, if not stated otherwise.

In by-visit summary tables only scheduled visits will be presented. All visits (both scheduled and unscheduled) will be presented in listings.

#### 7.2 Randomization and Blinding Process

This study is a randomized, double-blind, placebo-controlled study design. Patients will be randomized to treatment, either placebo or two different doses of SPI-1005 (1:1:1).

Study center and sponsor personnel involved in the conduct and interpretation of the study will not have access to treatment codes. Laboratory personnel, and contracted designees of SPI who statistically analyze the data, will be blinded to the study treatment received by each study participant. The bioanalytical staff analyzing PK samples will be provided a copy of the random codes but will not report unblinded data until after database lock. The sponsor's medical monitor will receive each treatment code in individual envelopes for use in emergency unblinding.

Apart from this, the data management and biostatistics team will be blinded until the database closure. The lead statistician will receive a copy of the unblinded treatment group after the database lock upon receiving a written authorization from the head of Biometrics/Statistics Lead from Sound Pharma to unblind the study.




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### 7.3 Analysis Population

#### 7.3.1 Randomized Population

The randomized population includes all patients who are randomized for treatments. Patients who have a missing randomization number will be included in this population. This includes patients who answer the question "Is the subject to be randomized?" = 'Yes" and with a non-missing "Subject Identification Code".

#### 7.3.2 Intent-to-Treat (ITT) Analysis Population

The ITT Efficacy Analysis population includes all patients from the randomized population who have received at least one dose of study drug and who have an evaluated post baseline efficacy assessment. The efficacy assessments include the evaluation of:

- Non- missing Pure-tone audiometry at Visit 3 or Visit 4
- Non- missing Words-in-Noise Test at Visit 3 or Visit 4
- Non- missing Tinnitus Functional Index (TFI) at Visit 2 or Visit 3 or Visit 4
- Non- missing Tinnitus Loudness (TL) at Visit 2 or Visit 3 or Visit 4
- Non- missing Vertigo Symptom Scale (VSS) at Visit 2 or Visit 3 or Visit 4

### 7.3.3 Safety Analysis Population

All study participants receiving at least one study treatment dose will be included in the safety analysis, whether or not they complete the study. The safety population is derived from the patients with evidence of receiving the study treatment in the "Drug Accountability" and eCRF form met with the following criteria:

- "Study Medication dispensed?" as 'Yes' and
- "Date of Dispensing" and
- The value entered for "Number of Capsules Taken" is greater than or equals 1 (missing values are excluded)

The safety population will be the primary population for the safety analysis. Analyses on the safety population will be based on actual treatment received.

# 7.3.4 Per-Protocol Population

The Per-Protocol Population includes all patients who receive study treatment and have efficacy parameters at Visit 3 and have no major protocol deviations.



Sponsor Name: Sound Pharmaceuticals, Inc.

Version No.: Final 1.0  Sponsor Nan

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

The major protocol deviations include:

- Treatment compliance of <80% and >120%
- Did not meet inclusion/exclusion criteria
- Baseline overall WINT score ≥ 2x Standard Deviations above the mean (rounded down to nearest integer)
- Major protocol deviations impacting the primary efficacy outcome measure.

### 7.3.5 PK Analysis Population

Statistical Analysis Plan

The PK analysis population includes all randomized patients performing PK evaluations, with the study medication compliance, and have a PK profile at all visits. The patients with major protocol deviations impacting PK results will be excluded from the analysis.

#### 7.4 Protocol Violation

Protocol deviations will be summarized by deviation category and treatment group. This analysis will be performed for all randomized patients.

#### 7.5 Data Handling

# 7.5.1 Imputation of Missing data

Imputation for missing values are not applicable.

### 7.6 Sample Size Calculation

120 male and female adults with probable or definitive Meniere's disease. This Phase 2b study (SPI-1005-251), is adequately powered to demonstrate a 50% improvement in a symptom of MD using the responder analysis detailed in below with 40 study participants per treatment group.

#### 7.7 Interim Analysis

There is no interim analysis planned for this study.




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### 7.8 Definitions and Derived Variables

For the statistical analysis, two different doses and placebo will be denoted according to the following table.

| Treatment | Label |
|-----------------------|-----------------|
| SPI-1005 po BID 200mg | SPI-1005 200 mg |
| SPI-1005 po BID 400mg | SPI-1005 400 mg |
| Placebo po BID | Placebo |

In the following table, the definitions and calculation of derived variables are summarised.

| Variable / Term | Definition / Way of calculation |
|---|---|
| Baseline | The last assessment on or before to the treatment start date. The most recent measurement prior to treatment start regardless of whether the measurement is collected at a scheduled or unscheduled visit will be considered for the baseline. |
| End of study | The date on which the last patient completes the last visit (includes follow-up visit). |
| BMI | Weight in kg / Height in m <sup>2</sup> |
| Treatment Start | The earliest date of 'date of drug dispense' (Date of dispensing) from Study Drug Dispensing and Drug Accountability eCRF form, where the patient has: • Answered 'Yes' to question, Study medication dispensed? And, • Recorded at least one capsule used for the question, 'Number of capsules taken' If the drug administration date is unavailable and only the last dose date of the patient is available, then the Randomization date will be considered as the treatment start date. |



Statistical Analysis Plan


NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

| Variable / Term | Definition / Way of calculation |
|---|---|
| | The treatment end date is taken from the field: |
| | 'Date of last study medication taken' from 'Study Completion or Early |
| | Termination' page. |
| Treatment End | If the 'Date of last study medication taken' is missing and there is evidence |
| | that the patient has taken the study medication, the last visit date will be |
| | considered as 'Treatment end date'. |
| | An adverse event (AE) will be considered as treatment-emergent if the time |
| Treatment Emergent | of onset is on or after the time of the first randomized study drug |
| AE (TEAE) | administration (treatment start date). |
| Duration of exposure | Treatment end date - treatment start date + 1, refer to section 8.2.1 in SAI for details |
| Treatment compliance | (Total number of capsules used/Total number of capsules to be taken) *100, refer to section 8.2.2 in SAP for details |
| Geo CV% | sqrt(exp(log SD)-1)*100 |

### 7.9 Statistical Software

All statistical analyses will be performed with SAS®, Version 9.2 or higher on a MS-Windows platform.

### 8 STATISTICAL ANALYSES

#### 8.1.1 Subject Disposition

The number of patients who have completed the study or early termination from the study and reasons for discontinuations will be grouped by treatment. The summary of patient disposition will be tabulated for all randomized, safety, ITT and PK analysis populations.

#### 8.1.2 Inclusion/Exclusion Criteria

The number and percentage of patients violating each inclusion/exclusion criterion will be presented by criterion. Violation of inclusion/exclusion criteria will be listed.




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

### 8.1.3 Demographic Data and Baseline Characteristics

Demographic characteristics include age, gender, ethnicity. Baseline characteristics include height, weight, BMI, TFI, VSS, PTA and WINT.

Frequency and percentage will be presented for gender, ethnicity. Descriptive statistics will be presented for age (years), height (cm), weight (Kg), BMI (kg/m²). These analyses will be performed for the Randomized, Safety, ITT and Per-Protocol populations.

Demographic and baseline characteristics will be presented in the by-patient listings. A data listing will be produced for the randomization details.

#### 8.1.4 Medical History

Medical history terms will be coded using MedDRA dictionary version 19.1.

Medical history will be summarized by MedDRA system organ class and preferred term for safety population. All medical history will be listed by patient and treatment group.

### 8.1.5 Prior and Concomitant Medication

Prior and concomitant medications will be assessed at screening and at each subsequent study visit. Medications will be coded using WHO Drug Dictionary version MAR2017.

Medication will be classified as prior, if the end date is known and is before the first use of the study medication. Medications that are ongoing or ended after the first use of the study medication will be classified as concomitant. If the end date of the medication is unknown, it will also be considered concomitant. If the end date is partially known, the medication will be considered concomitant, unless the known part of the end date rules out the possibility that the medication could have ended before the start of the study drug.

Prior and concomitant medications will be separately summarized by ATC class (the highest available level) and preferred name for the safety population. The prior and concomitant medications will be listed in a by-patient listing.




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### 8.2 Extent of Exposure and Compliance

# **8.2.1** Treatment Exposure

Treatments will be dispensed at baseline to patients based on the randomized group assignments and the patients will receive the treatment for a duration of 28 days.

The earliest date of 'date of drug dispense' (Date of dispensing) from Study Drug Dispensing and Drug Accountability eCRF form, where the patient has:

- Answered 'Yes' to question, 'Study medication dispensed?' and,
- Recorded at least one capsule used for the question, 'Number of capsules taken'

If the drug administration date is unavailable and the last dose date of the patient is only available, then the Randomization date will be considered as treatment start date.

The treatment end date is taken from the field:

- 'Date of last study medication taken' from 'Study Completion or Early Termination' page. If the date of last study drug administration is missing and there is evidence that the patient has taken study medication, last visit date will be considered as 'Treatment end date'.
- Duration of treatment exposure is derived as treatment end date treatment start date + 1

The duration of treatment exposure will be summarized descriptively by treatment group for safety population. Data listing will be presented for study drug administration.

#### **8.2.2** Treatment Compliance

Treatment compliance is defined as intake of 80% to 120% of the dispensed capsules by an individual patient during the treatment period. Hence the compliance is computed as:

• (Total number of capsules used/Total number of capsules to be taken) \*100

Where the total number of capsules used is derived as the sum of results recorded for the question 'Number of capsules taken' in the drug accountability form.

Data listing also will be presented for treatment compliance.

### 8.3 Efficacy Analysis

#### 8.3.1 Analysis of Primary Endpoint

Primary analyses will use the Per-Protocol analysis population and Intent-To-Treat analysis population.




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### **8.3.1.1** Pure-Tone Audiometry

Pure-tone audiometry (PTA) will be measured at visit 1, visit 3 and visit 4.

Both the actual ear value and calculated change from baseline PTA data will be summarized by visits and treatment groups.

PTA data will be analyzed with a mixed-effects model for repeated measures, and a post-hoc Bonferroni correction analysis with significance set to 0.05. The calculated change of PTA data will be calculated by the difference of the actual ear value at baseline and the actual ear value at each visit post baseline. The primary assessment of PTA data will consider a  $\geq$ 10 dBHL improvement from baseline as a clinically relevant response (only low frequency: 250, 500, 1000 Hz). The secondary assessments of PTA data will consider an improvement from baseline of  $\geq$ 10 dBHL at two adjacent frequencies or  $\geq$ 20 dBHL at one frequency as clinically relevant responses (only low frequency: 250, 500, 1000 Hz). The final processed data will be analyzed using a chi-square test or Fisher's Exact test to assess the improvement between treatment groups.

#### 8.3.1.2 Words-in-Noise Test

The Words-in-Noise Test (WINT) will be measured at visit 1, visit 3 and visit 4.

Both the actual ear value and calculated change from baseline WINT data will be summarized by visits and treatment groups.

WINT data will be analyzed with a mixed-effects model for repeated measures, and a post-hoc Bonferroni correction analysis with significance set to 0.05. The calculated change of WINT data will be calculated by the difference of the actual ear value at baseline and the actual ear result at each visit post baseline. The primary assessment of WINT data will consider a  $\geq 10\%$  improvement from baseline as a clinically relevant response. The secondary assessments of WINT data will consider an improvement from baseline of  $\geq 20\%$  or  $\geq 4$  words as clinically relevant responses. The final processed data will be analyzed using a chi-square test or Fisher's Exact test to assess the improvement between treatment groups.

#### 8.3.1.3 Tinnitus Functional Index (TFI)

The Tinnitus Functional Index (TFI) will be measured at visit 1, visit 2, visit 3 and visit 4.

The actual patient reported outcome (PRO) value and change from baseline TFI will be summarized by visits and treatment groups.

TFI will be analyzed as a composite score and for the following individual subscales: Intrusiveness, Sense of control, Cognition, Sleep, Auditory, Relaxation, Quality of life, and Emotional.




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

The overall total score will be calculated by the sum of all valid answers from both TFI pages and will be divided by the number of questions for which that respondent provided valid answers and then multiplied by 10.

| SUBSCALE NAME | ITEMS IN SUBSCALE |
|-----------------------|--------------------|
| INTRUSIVE | #1, #2, #3 |
| SENSE OF CONTROL | #4, #5, #6 |
| COGNITIVE | #7, #8, #9 |
| SLEEP | #10, #11, #12 |
| AUDITORY | #13, #14, #15 |
| RELAXATION | #16, #17, #18 |
| QUALITY OF LIFE (QOL) | #19, #20, #28, #22 |
| EMOTIONAL | #23, #24, #25 |

Each of the 8 subscales consists of 3 items (except for the Quality of life subscale, which consists of 4 items). For subscale scores to be valid no more than 1 item should be omitted. Computation of subscale scores is calculated as:

- 1) Sum all respondent's valid answers for a given subscale.
- 2) Divide that number by the number of valid answers that were provided by that respondent for that subscale.
- 3) Multiply by 10. For the respondent in question, this procedure generates a subscale score in the range 0-100 for each valid subscale.

Overall TFI score is not valid if the respondent omits seven or more items. To be considered a valid measure of tinnitus severity, the respondent must answer at least 19 items.

The TFI data will be analyzed with a mixed-effects model for repeated measures, and a post-hoc Bonferroni correction analysis with significance set to 0.05. The calculated change of TFI data will be calculated as the difference of the PRO value at baseline and the PRO value at each post baseline timepoint. The improvement will be considered only if the difference between post baseline and baseline value is  $\geq$ 10 pts. The final processed data will be analyzed using a chi-square test or Fisher's Exact test to assess the improvement between treatment groups.




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### **8.3.1.4** Tinnitus Loudness

Tinnitus loudness (TL) will be measured at visit 1, visit 2, visit 3 and visit 4. TL is assessed from question number two of the TFI.

The actual patient reported outcome (PRO) value and change from baseline for TL will be summarized by visits and treatment groups. TL data will be analyzed with a mixed-effects model for repeated measures, and a post-hoc Bonferroni correction analysis with significance set to 0.05. The calculated change of TL data will be calculated as the difference of the PRO value at baseline and the PRO value at each post baseline timepoint. The improvement will be considered only if the difference between post baseline and baseline value is  $\geq 2$  pts. The final processed data will be analyzed using a chi-square test or Fisher's Exact test to assess the improvement between treatment groups.

### 8.3.1.5 Vertigo Symptom Scale

Vertigo Symptom Scale (VSS) will be measured at visit 1, visit 2, visit 3 and visit 4.

The actual patient reported outcome (PRO) value and change from baseline for VSS will be summarized by visits and treatment groups.

VSS will be analyzed for Total Scale, Vertigo/balance sub-scale and Autonomic/anxiety sub-scale. The Vertigo/balance sub-scale will be calculated as the sum of questions 1, 3, 4, 6, 8, 10, 13 and 15. The Autonomic/anxiety sub-scale will be calculated as the sum of questions 2, 5, 7, 9, 11, 12 and 14. The range for the Vertigo/balance sub-scale will be 0-32 and the range for Autonomic/anxiety sub-scale will be 0-28.

VSS data will be analyzed with a mixed-effects model for repeated measures, and a post-hoc Bonferroni correction analysis with significance set to 0.05.

The calculated change of VSS data will be calculated as the difference of the PRO value at baseline and the PRO value at each post baseline timepoint. The improvement will be considered only if the difference between post baseline and baseline value is  $\geq 6$  pts. The final processed data will be analyzed using a chi-square test or Fisher's Exact test to assess the improvement between treatment groups.



Version No.: Final 1.0 

Sponsor Study No: SPI-1005-251

Sponsor Name: Sound Pharmaceuticals, Inc.

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### 8.4 Safety Analysis

#### **8.4.1** Adverse Events

Adverse Events will be coded using the Medical Dictionary of Regulatory Activities (MedDRA version 19.1), the coded terms will be used for summarizing the AE(s).

An AE will be considered as treatment-emergent if the time of onset is on or after the time of the first randomized study drug administration. AEs with unknown start dates will be counted as treatment-emergent unless the AE resolution date is prior to the study drug start date. If the start date is partially missing, AE will be considered treatment-emergent unless the known part of the start date or the end date rules out that it occurred after the start of the study drug.

An overall summary table which summarizes, the number and percentages of patients with adverse events, treatment emergent adverse events, serious adverse events, adverse events leading to death and adverse events related to study drug will be provided by treatment groups.

Patients experiencing any adverse events will be summarized by Preferred Term (PT), SOC and treatment. Furthermore, listings of SAEs and AEs that lead to withdrawal will be provided. The number and percentage of patients with at least one TEAE, SAE and discontinuation of study treatment due to AE (DAE) will be summarized by system organ class, preferred term and treatment group.

Adverse Events will be summarized by System Organ Class, Preferred Term and Treatment for Any Adverse Events, Serious Adverse Events, Adverse Events leading to medication discontinuation, Adverse leading to death, Adverse Events by severity, Adverse Events by outcome and Adverse Events by relationship.

A patient experiencing the same AE multiple times will be counted only once for that preferred term. Similarly, if a patient experiences multiple AEs within the same system organ class that patient will be counted only once in that system organ class. In summaries by severity or by relationship, if a patient has the same AE on multiple occasions, the highest severity, and the closest relationship to study drug, respectively, will be used for summary.

All information pertaining to adverse events noted during the study regardless of treatment emergent or not will be listed by patient, detailing verbatim, preferred term, system organ class, start date, stop date, TEAE status, severity, outcome, action taken and causal relationship to the study drug.



Statistical Analysis Plan


NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### 8.4.2 Clinical Laboratory Evaluations

Blood samples for clinical safety laboratory assessments will be collected at the following time Visit 1, Visit 2, Visit 3 and Visit 4. The following parameters will be analyzed under these categories:

| Hematology | Chemistry | |
|-------------|--------------------------------------|----------------------|
| RBC | Sodium | Albumin |
| Hematocrit | Potassium | AST (SGOT) |
| Hemoglobin | Chloride | ALT (SGPT) |
| Platelets | Bicarbonate | GGT |
| WBC | Glucose | Total bilirubin |
| Neutrophils | Blood urea nitrogen<br>(BUN) or Urea | Alkaline phosphatase |
| Lymphocytes | Creatinine | Uric acid |
| Monocytes | Calcium | LDH |
| Basophils | Magnesium | Cholesterol |
| Eosinophils | Inorganic phosphorus | Triglycerides |
| | Total protein | |

Laboratory results will be summarized descriptively for actual and change from baseline values by visits and treatment for each category of clinical chemistry and hematology. In addition, baseline shift tables will be presented for the lab parameters by visits and treatments for laboratory categories, the results falling out of normal ranges will be classified as Normal, Abnormal High and Abnormal Low and will be used for the shift tables. The 'Normal', 'Abnormal Low' and 'Abnormal High' values are determined based on the laboratory normal ranges. The number and percentage of patients reaching 'Normal', 'Abnormal CS' and 'Abnormal NCS' results for laboratory parameters will be summarized All laboratory results will be listed in data listings, the abnormal values will be flagged in the listings.



Version No.: Final 1.0 

Sponsor Study No: SPI-1005-251

Sponsor Name: Sound Pharmaceuticals, Inc.

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### 8.4.3 Vital Signs

Vital signs will be measured at Visit 1, Visit 2, Visit 3 and Visit 4.

The vital signs parameters include:

- Systolic Blood Pressure (mmHg)
- Diastolic Blood Pressure (mmHg)
- Pulse Rate (Beats/min)
- Oral Temperature (°C)

The actual and change from baseline vital signs parameters will be summarized descriptively by visits and treatment groups.

In addition, number and percentage of patients reaching 'Normal', 'Abnormal CS' and 'Abnormal NCS' results for vital signs parameters will be summarized by visits and treatment groups. Data listings will be presented for vital signs parameters.

Shift tables for the overall interpretation of vital signs parameters will be summarized by visits and treatment groups.

# 8.4.4 Physical examination

Physical examination will be performed at Visit 1, Visit 2, Visit 3 and Visit 4. Physical examination will include an examination of skin, HEENT (Otoscopic exam) Head/ Eyes/ Ears/Nose/Throat/Thyroid, Respiratory, Cardiovascular, Abdomen, Musculoskeletal, Neurological (and reflexes), Gastrointestinal, Endocrine, Lymph nodes and others.

A summary of these findings, number and percentages of patients achieving 'Normal', 'Abnormal CS', 'Abnormal NCS' will be presented by visit, body system and treatment group. Results will also be listed.

#### 8.5 Pharmacokinetic Analysis

The PK analysis will be performed based on PK analysis population.

Three (3) mL of blood will be collected at visit 1, visit 2, visit 3 and visit 4. Study participants should be instructed to refrain from taking their morning dose until after their blood is drawn at Clinic Visit 2 and Clinic Visit 3. Sample collection times (actual clock time using 24:00) are to be recorded and will be captured in the CRF.



 Sponsor Name: Sound Pharmaceuticals, Inc.

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

The patient listings as well as Patient's PK profile plots in actual and semi-logarithmic views will be prepared for the PK concentrations. Descriptive summary statistics table including geometric mean & CV% geometric mean will be presented by timepoints and treatment groups. In addition, mean  $\pm$  SD graphs will be prepared for the concentration by timepoints and treatment groups.

Descriptive statistics including geometric mean & CV% geometric mean will be presented for the PK parameters, AUC  $_{0\text{-t}}$  (mg. h/L) and  $C_{max}$  (mg/L).

### 8.6 Multicentre Studies

Statistical Analysis Plan

Version No.: Final 1.0

Patients from thirteen sites in U.S. participated in the study and all the data across the sites will be presented.

### 8.7 Subgroup Analyses

Not Applicable




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

# 9 DEVIATION FROM THE STUDY PROTOCOL

The differences between study protocol and statistical analysis plan are summarised in the following table:

| Change | Study Protocol | Statistical Analysis Plan |
|---|---|---|
| 6.2 Study | The primary objective of this | > To determine the Safety of SPI-1005 |
| Objectives | Phase 2 study is to determine the: | treatment in adults with Meniere's |
| | <ul> <li>Safety of SPI-1005</li> </ul> | disease. |
| | treatment in adults with | ➤ To determine the Efficacy of SPI- |
| | Meniere's disease. | 1005 with the following clinically |
| | • Efficacy of SPI-1005 will | validated methods and measures |
| | be determined by the | (responder analysis): |
| | - | <ul> <li>Primary pure-tone</li> </ul> |
| | following | audiometry assessment: |
| | clinically significant methods and | (250, 500 or 1000 Hz): |
| | measures (responder | Improvements from baseline |
| | analysis): | of ≥10 dB Secondary pure- |
| | ■ Pure tone | tone audiometry assessments |
| | audiometry (>30 | (250, 500 or 1000 Hz): |
| | dBHL at 250, 500 | Improvements from baseline |
| | or 1000 Hz) | of ≥10 dB at 2 frequencies or |
| | >10 dB | ≥20 dB at 1 frequency |
| | improvement from | ■ Primary Words-in-Noise |
| | baseline | Test assessment (0-35): |
| | ■ Words in Noise | Improvements from baseline |
| | | of≥10% |
| | Test (0-35) | <ul> <li>Secondary Words-in-Noise</li> </ul> |
| | >10 % increase | Test assessments (0-35): |
| | from baseline | Improvements from baseline |
| | ■ Tinnitus | of ≥20% or ≥4 words |
| | Functional Index | Tinnitus Functional Index |
| | (TFI) (0-100) | $(TFI): (0-100) \ge 10 \text{ pt.}$ |
| | | reduction from baseline |



Statistical Analysis Plan


NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

>10 pt. reduction from baseline

- Tinnitus
   Loudness: Q#2 of
   TFI (0-10)
   >2 pt. reduction
   from baseline
- Vertigo SymptomScale (0-60)>6 pt. reductionfrom baseline

The responder analysis from each method and measure will be compared between treatment groups for significance.

- Efficacy of SPI-1005 treatment in adults with Meniere's disease based on
- Improvement in sensorineural hearing loss using pure tone audiometry at 250, 500, or 1000 Hz; or
- Word recognition score using WIN testing at 24, 20,16, 12, 8, 4 and 0 SNR; or

- Tinnitus Loudness: Q#2 of TFI: (0-10) ≥ 2 pt. reduction from baseline
- Vertigo Symptom Scale
   (0-60): ≥ 6 pt. reduction
   from baseline

The responder analysis from each method and measure will be compared between treatment groups for significance.

- The efficacy of SPI-1005 treatment in adults with Meniere's disease will be based on:
  - Improvement in sensorineural hearing loss using pure tone audiometry at 250, 500, or 1000 Hz; or
  - ➤ Word recognition score using WINT at 24, 20,16, 12, 8, 4 and 0 SNR; or
  - ➤ Improvement in the Tinnitus Functional Index (TFI); or
  - Improvement in Tinnitus Loudness (TL); or
  - > Improvement in the Vertigo Symptoms Scale (VSS)

# 9.1.1 Exploratory Analysis

Primary pure-tone audiometry assessment: (250, 500 or 1000 Hz):
 Improvements from baseline of ≥10 dB




Secondary pure-tone audiometry Improvement in assessments (250, 500 or 1000 the Tinnitus Improvements Hz): from Functional Index baseline of  $\geq 10$  dB at 2 (TFI); or frequencies or  $\geq 20$  dB at 1 Improvement in frequency Tinnitus Loudness ■ Primary Words-in-Noise Test (TL); or assessment (0-35): Improvements Improvement in from baseline of  $\geq 10\%$ the Vertigo Secondary Words-in-Noise Test Symptoms Scale assessments (0-35): Improvements (VSS). from baseline of  $\geq 20\%$  or  $\geq 4$  words The secondary objectives of this study are to determine the: • Pharmacokinetics of SPI-1005.

# 10 SOPS FOR ANALYSIS AND REPORTING

Ecron Acunova's standard operating procedures as well as the ICH guideline E9 will be applied to this analysis. The structure of post-text-tables and the appendices will be in accordance with the ICH guideline E3.

# 11 DATABASE LOCK AND UNBLINDING

After the data cleaning process is finalised according to the data management manual and the assignment of patients to the analysis population is agreed and signed by the sponsor, the data base will be locked. SAS datasets will be extracted from the data.

After the data base closure, unblinding of randomization will be initiated and the randomisation dataset will be prepared, and it will be validated by a second person.

#### **Confidentiality Statement**

This document is confidential and proprietary to Sponsor and EA and for restricted circulation and access only. No part of it may be transmitted, reproduced, published or used by any person/s without prior written authorization.



Sponsor Name: Sound Pharmaceuticals, Inc. Version No.: Final 1.0 

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### 12 **REFERENCES**

Further references are given in the study protocol.



Sponsor Name: Sound Pharmaceuticals, Inc. Version No.: Final 1.0 

NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

#### 13 LIST OF REPORTED TABLES

| Table No. | Table |
|---|---|
| 14.1 | Demography Analysis |
| TABLE 14.1.1 | Summary of Patient Disposition (Randomized Population) |
| TABLE 14.1.1.1 | Summary of Patient Disposition (Safety Population) |
| TABLE 14.1.1.2 | Summary of Patient Disposition (Intent-to-Treat Population) |
| TABLE 14.1.1.3 | Summary of Patient Disposition (Per-Protocol Population) |
| TABLE 14.1.2 | Summary of Eligibility Status (All Screened Subjects) |
| TABLE 14.1.3 | Number of Patient Included and Excluded from Analysis Population |
| TABLE 14.1.4 | Reason for Patient Excluded from Analysis Population (Randomized Population) |
| TABLE 14.1.5 | Summary of Protocol Deviations (Randomized Population) |
| TABLE 14.1.6 | Number of Patient at Each Visit (Randomized Population) |
| TABLE 14.1.7 | Number of Patient Enrolled by Study Center (Randomized Population) |
| TABLE 14.1.8 | Summary of Patient Demographic Characteristics at Baseline (Randomized Population) |
| TABLE 14.1.8.1 | Summary of Patient Demographic Characteristics at Baseline (Safety Population) |
| TABLE 14.1.8.2 | Summary of Patient Demographic Characteristics at Baseline (Intent-to-Treat Population) |
| TABLE 14.1.8.3 | Summary of Patient Demographic Characteristics at Baseline (Per-Protocol Population) |
| TABLE 14.1.9 | Summary of Medical History Classified by MedDRA Preferred Term (Safety Population) |
| TABLE 14.1.10 | Summary of Prior Medications by ATC Class and Preferred Term (Safety Population) |
| TABLE 14.1.11 | Summary of Concomitant Medication by ATC Class and Preferred Term (Safety Population) |
| TABLE 14.1.12 | Summary of Study Treatment Taken by the Patient: (Safety Population) |
| 14.2 | Efficacy Analysis |
| TABLE 14.2.1 | Summary and Analysis of Actual and Change from Baseline of Pure-Tone Audiometry(PTA) – Continuous variable (Intent-to-Treat Population) |




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

| Table No. | Table |
|---|---|
| TABLE 14.2.1.1 | Summary and Analysis of Actual and Change from Baseline of Pure-<br>Tone Audiometry(PTA) – Continuous variable (Per-Protocol Population) |
| TABLE 14.2.1.2 | Post-hoc analysis for Pure-Tone Audiometry (PTA) (Intent-to-Treat Population) |
| TABLE 14.2.1.3 | Post-hoc analysis for Pure-Tone Audiometry (PTA) (Per-Protocol Population) |
| TABLE 14.2.1.4 | Summary and Analysis of Pure- Tone Audiometry(PTA) >=10 DB improvement from Baseline (Intent-to-Treat Population) |
| TABLE 14.2.1.5 | Summary and Analysis of Pure- Tone Audiometry(PTA) >=10 DB improvement from Baseline (Per-Protocol Population) |
| TABLE 14.2.1.6 | Summary and Analysis for Pure-Tone Audiometry (PTA) ≥10 dB Improvement from Baseline atleast 2 Frequencies (Intent-to-Treat Population) |
| TABLE 14.2.1.7 | Summary and Analysis for Pure-Tone Audiometry (PTA) ≥10 dB Improvement from Baseline atleast 2 Frequencies (Per-Protocol Population) |
| TABLE 14.2.1.8 | Summary and Analysis for Pure-Tone Audiometry (PTA) ≥20 dB Improvement from Baseline atleast 1 Frequency (Intent-to-Treat Population) |
| TABLE 14.2.1.9 | Summary and Analysis for Pure-Tone Audiometry (PTA) ≥20 dB Improvement from Baseline atleast 1 Frequency (Per-Protocol Population) |
| TABLE 14.2.2 | Summary and Analysis of Actual and Change from Baseline of Words-in-<br>Noise Test(WINT) – Continuous Variable (Intent-to-Treat Population) |
| TABLE 14.2.2.1 | Summary and Analysis of Actual and Change from Baseline of Words-in-<br>Noise Test (WINT) – Continuous Variable (Per-Protocol Population) |
| TABLE 14.2.2.2 | Post-hoc analysis for Words-in-Noise Test (WINT) (Intent-to-Treat Population) |
| TABLE 14.2.2.3 | Post-hoc analysis for Words-in-Noise Test (WINT) (Per-Protocol Population) |
| TABLE 14.2.2.4 | Summary and Analysis Words-in-Noise Test(WINT) >=10% Increase from Baseline (Intent-to-Treat Population) |
| TABLE 14.2.2.5 | Summary and Analysis of Words-in-Noise Test(WINT) >=10% Increase from Baseline (Per-Protocol Population) |
| TABLE 14.2.2.6 | Summary and Analysis for Words-in-Noise Test (WINT) ≥20% Increase from Baseline (Intent-to-Treat Population) |
| TABLE 14.2.2.7 | Summary and Analysis for Words-in-Noise Test (WINT) ≥20% Increase from Baseline (Per-Protocol Population) |




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

| Table No. | Table |
|---|---|
| TABLE 14.2.2.8 | Summary and Analysis for Words-in-Noise Test (WINT) ≥ 4 Words Increase from Baseline (Intent-to-Treat Population) |
| TABLE 14.2.2.9 | Summary and Analysis for Words-in-Noise Test (WINT) ≥ 4 Words Increase from Baseline (Per-Protocol Population) |
| TABLE 14.2.3 | Summary and Analysis of Actual and Change from Baseline of Tinnitus Functional Index (TFI) – Continuous Variable (Intent-to-Treat Population) |
| TABLE 14.2.3.1 | Summary and Analysis of Actual and Change from Baseline of Tinnitus<br>Functional Index (TFI) – Continuous Variable (Per-Protocol Population) |
| TABLE 14.2.3.2 | Post-hoc analysis for Tinnitus Functional Index (TFI) (Intent-to-Treat Population) |
| TABLE 14.2.3.3: | Post-hoc analysis for Tinnitus Functional Index (TFI) (Per-Protocol Population) |
| TABLE 14.2.3.4 | Summary and Analysis of Tinnitus Functional Index (TFI) ≥ 10pt. reduction from Baseline (Intent-to-Treat Population) |
| TABLE 14.2.3.5 | Summary and Analysis of Tinnitus Functional Index (TFI) ≥ 10pt. reduction from Baseline (Per-Protocol Population) |
| TABLE 14.2.4 | Summary and Analysis of Actual and Change from Baseline of Tinnitus Loudness(TL) – Continuous Variable (Intent-to-Treat Population) |
| TABLE 14.2.4.1 | Summary and Analysis of Actual and Change from Baseline of Tinnitus Loudness (TL) – Continuous Variable (Per-Protocol Population) |
| TABLE 14.2.4.2 | Post-hoc analysis for Tinnitus Loudness (TL) (Intent-to-Treat Population) |
| TABLE 14.2.4.3 | Post-hoc analysis for Tinnitus Loudness (TL) (Per-Protocol Population) |
| TABLE 14.2.4.4 | Summary and Analysis of Tinnitus Loudness (TL) $\geq$ 2pt. reduction from Baseline (Intent-to-Treat Population) |
| TABLE 14.2.4.5 | Summary and Analysis of Tinnitus Loudness (TL) $\geq$ 2pt. reduction from Baseline (Per-Protocol Population) |
| TABLE 14.2.5 | Summary and Analysis of Actual and Change from Baseline of Vertigo Symptom Scale (VSS) – Continuous Variable (Intent-to-Treat Population) |
| TABLE 14.2.5.1 | Summary and Analysis of Actual and Change from Baseline of Vertigo<br>Symptom Scale (VSS) – Continuous Variable (Per-Protocol Population) |
| TABLE 14.2.5.2 | Post-hoc analysis for Vertigo Symptom Scale (VSS) (Intent-to-Treat Population) |
| TABLE 14.2.5.3 | Post-hoc analysis for Vertigo Symptom Scale (VSS) (Per-Protocol Population) |




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

| Table No. | Table |
|---|---|
| TABLE 14.2.5.4 | Summary and Analysis of Vertigo Symptom Scale (VSS) ≥ 6pt. reduction from Baseline (Intent-to-Treat Population) |
| TABLE 14.2.5.5 | Summary and Analysis of Vertigo Symptom Scale (VSS) ≥ 6pt. reduction from Baseline (Per-Protocol Population) |
| TABLE 14.2.6 | Summary of PK Concentration values (PK Population) |
| TABLE 14.2.7 | Summary of PK parameters by (PK Population) |
| 14.3 | Safety Analysis |
| TABLE 14.3.1 | Overall Summary of Adverse Events (Safety Population) |
| TABLE 14.3.2 | Number (and Percentage) of Patient with Adverse Events Classified by<br>System Organ Class, Preferred Term During The Study (Safety<br>Population) |
| TABLE 14.3.2.1 | Number (and Percentage) of Patient with Adverse Events Classified by<br>Treatment Emergent Adverse Events (Safety Population) |
| TABLE 14.3.2.2 | Number (and Percentage) of Patient Discontinuation of Study Treatment<br>Due to AE Classified by System Organ Class, Preferred Term During The<br>Study (Safety Population) |
| TABLE 14.3.2.3 | Number (and Percentage) of Patient Death Classified by System Organ Class, Preferred Term During The Study (Safety Population) |
| TABLE 14.3.3 | Number (and Percentage) of Patient with Adverse Events Classified by Severity (Safety Population) |
| TABLE 14.3.4 | Number (and Percentage) of Patient with Adverse Events Classified by<br>System Organ Class, Preferred Term and Relation to Study Medication<br>(Safety Population) |
| TABLE 14.3.5 | Number (and Percentage) of Patient With Adverse Events Classified by Action taken with Study Drug (Safety Population) |
| TABLE 14.3.6 | Number (and Percentage) of Patient with Adverse Events Classified Outcome (Safety Population) |
| TABLE 14.3.7 | Number (and Percentage) of Patient With Serious Adverse Events System<br>Organ Class and Preferred Term (Safety Population) |
| TABLE 14.3.8 | Summary of Physical Examination by Visit (Safety Population) |
| TABLE 14.3.9 | Summary of Actual and Change from Baseline for Vital Signs by Visit:<br>Continuous Variable (Safety Population) |
| TABLE 14.3.10 | Summary of Vital Signs by Visit: Categorical Variable (Safety Population) |




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

| Table No. | Table |
|---|---|
| TABLE 14.3.11 | Summary of Shift from Baseline of Vital Signs by Visit: Categorical Variable (Safety Population) |
| TABLE 14.3.12 | Summary and Change from Baseline of Lab parameters(Hematology) by Visit and Treatment (Safety Population) |
| TABLE 14.3.13 | Summary and Change from Baseline Lab Parameters (Clinical Chemistry) by Visit and Treatment (Safety Population) |
| TABLE 14.3.14 | Summary of Shift from Baseline of Lab Parameter (Hemotology) Results Based on the Reference Range by Visit and Treatment: Categorical Variable (Safety Population) |
| TABLE 14.3.15 | Summary of Shift from Baseline of Lab Parameter (Hemotology) Results Based on the Reference Range by Visit and Treatment: Categorical Variable (Safety Population) |
| TABLE 14.3.16 | Summary of Lab Parameters (Urine Pregnancy) (Point of care testing) by Treatment (Safety Population) |



Statistical Analysis Plan


NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

# 14 LIST OF REPORTED FIGURES

- 15.1 Mean (± SD) Graph for Pure Tone Audiometry (PTA) (Intent to Treat Population)
  - 15.1.1 Mean (± SD) Graph for Pure Tone Audiometry (PTA) (Per-Protocol Population)
  - 15.2 Mean (± SD) Graph for Words in Noise Test (WINT) (Intent-to-Treat Population)
  - 15.2.1 Mean (± SD) Graph for Words in Noise Test (WINT) (Per-Protocol Population)
  - 15.3 Mean (± SD) Graph for Tinnitus Functional Index (TFI) (Intent-to-Treat Population)
  - 15.3.1 Mean (± SD) Graph for Tinnitus Functional Index (TFI) (Per-Protocol Population)
  - 15.4 Mean (± SD) Graph for Mean (± SD) Graph for Tinnitus Loudness(Intent-to-Treat Population)
  - 15.4.1 Mean (± SD) Graph for Tinnitus Loudness (Per-Protocol Population)
  - 15.5 Mean (± SD) Graph for Vertigo Symptom Scale(Intent-to-Treat Population)
  - 15.5.1 Mean (± SD) Graph for Vertigo Symptom Scale (Per-Protocol Population)
  - 15.6 Graph for Pure-tone audiometry ≥10 dB improvement from baseline (Intent-to-Treat Population)
  - 15.6.1 Graph for Pure-tone audiometry ≥10 dB improvement from baseline (Per-Protocol Population)
  - 15.6.2 Graph for Words-in-Noise Test ≥10% increase from baseline (Intent-to-Treat Population)
  - 15.6.3 Graph for Words-in-Noise Test ≥10% increase from baseline (Per-Protocol Population)
  - 15.6.4 Graph for Tinnitus Functional Index (TFI) ≥10 pt. Reduction from baseline (Intent-to-Treat Population)
  - 15.6.5 Graph for Tinnitus Functional Index (TFI) ≥10 pt. Reduction from baseline (Per-Protocol Population)
  - 15.6.6 Graph for Tinnitus Loudness ≥2 pt Reduction from baseline (Intent-to-Treat Population)
  - 15.6.7 Graph for Tinnitus Loudness ≥2 pt Reduction from baseline (Per-Protocol Population)
  - 15.6.8 Graph for Vertigo Symptom Scale ≥6 pt. Reduction from baseline (Intent-to-Treat Population)
  - 15.6.9 Graph for Vertigo Symptom Scale ≥6 pt. Reduction from baseline (Per-Protocol Population)
  - 15.6.10 Graph for Pure-Tone Audiometry (PTA)≥10 dB Improvement from Baseline at 2 Frequencies (Intent-to-Treat Population)
  - 15.6.11 Graph for Pure-Tone Audiometry (PTA) ≥10 dB Improvement from Baseline at 2 Frequencies (Per-Protocol Population)
  - 15.6.12 Graph for Pure-Tone Audiometry (PTA) ≥20 dB Improvement from Baseline at 1 Frequency (Intent-to-Treat Population)
  - 15.6.13 Graph for Pure-Tone Audiometry (PTA) ≥20 dB Improvement from Baseline at 1 Frequency (Per-Protocol Population)




NLS Study Code: SPI-1005-251 Short Title of Study: SPI-1005-251 (Sound Pharmaceuticals, Inc)

15.6.14 Graph for Words-in-Noise Test (WINT) ≥20% Increase from Baseline (Intent-to-Treat Population)

- 15.6.15 Graph for Words-in-Noise Test (WINT) ≥20% Increase from Baseline (Per-Protocol Population)
- 15.6.16 Graph for Words-in-Noise Test (WINT) >= 4 Words Increase from Baseline (Intent-to-Treat Population)
- 15.6.17 Graph for Words-in-Noise Test (WINT) >= 4 Words Increase from Baseline (Per-Protocol Population)
- 15.7 Individual Profile Graph for PK Concentration (PK Population)
- 15.8 Mean Graph for PK Concentration (PK Population)




NLS Study Code: SPI-1005-251

Short Title of Study: SPI -1005 -251 (Sound Pharmaceuticals, Inc)

# 15 LIST OF REPORTED SUBJECT DATA LISTINGS

- 16.2.1 Discontinued Patient
  - 16.2.1.1 Inclusion / Exclusion Criteria
  - 16.2.1.2 Randomization
  - 16.2.1.3 Protocol Violations
- 16.2.2 Patient excluded from the analysis
  - 16.2.2.1 Patient Excluded from the Analysis population
  - 16.2.2.2 Comments
- 16.2.3 Demographic and baseline data
  - 16.2.3.1 Patient Demographic, Exposure and Disposition
  - 16.2.3.2 Medical History
  - 16.2.3.3 Prior/Concomitant Medications
- 16.2.4 Compliance
  - 16.2.4.1 Study Drug Administration, Accounting and Compliance
- 16.2.5 Individual efficacy response data
  - 16.2.5.1 Tinnitus Functional Index Results
  - 16.2.5.2 Vertigo Symptom Scale(VSS) Scores Results
  - 16.2.5.3 Words-in-Noise Test Results (WINT)
  - 16.2.5.4 Pure-tone audiometry Results-Air Conduction(dB)
  - 16.2.5.5 Pure-tone audiometry Results-Bone Conduction(dB)
  - 16.2.5.6 PK Sampling
  - 16.2.5.7 PK Parameters
- 16.2.6 Adverse event
  - 16.2.6.1 Patient Adverse Event
- 16.2.7 Listing of Individual Lab Measurements by Patient
  - 16.2.7.1 Clinical Lab Results
  - 16.2.7.2 Vital Signs
  - 16.2.7.3 Physical Examination